CLINICAL TRIAL: NCT02046187
Title: Phase I/II Prospective Trial for Newly Diagnosed GBM, With Upfront Gross or Subtotal Resection, Followed by Ketogenic Diet With Radiotherapy and Concurrent Temodar(R) Chemotherapy Followed by Adjuvant Temodar(R) Chemotherapy.
Brief Title: Ketogenic Diet With Radiation and Chemotherapy for Newly Diagnosed Glioblastoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: excessive protocol deviations due to strict nature of diet requirements
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KD-13BN069
Record Dates: First submitted 2014-01-17; First posted 2014-01-27 (Estimated); Last update posted 2021-06-16 (Actual); Status verified 2021-06

CONDITIONS: Glioblastoma (GBM)
Keywords: Ketogenic Diet; Brain tumor; Glioma; Glioblastoma; Radiation; Chemotherapy; temozolomide
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms; Glioma | interventions — Diet, Ketogenic; Radiotherapy; Temozolomide; Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ketogenic Diet (Experimental): Subjects will adhere to a ketogenic diet prior to the start of and through radiation therapy course until the time of first scan after radiation ends. During radiation course, patients also take temozolomide daily.
  Interventions: Dietary Supplement: Ketogenic Diet; Radiation: Radiation therapy; Drug: Temozolomide

INTERVENTIONS:
Dietary Supplement: Ketogenic Diet — Patients/families meet with the study dietician after surgery to discuss the ketogenic diet (KD), ask questions and plan clinic visits. Before radiation and chemotherapy begins, training takes place about the diet, meal planning and ketone/glucose monitoring. Ketosis will begin with the help of the dietitian one week before radiation begins. The patient will follow a classic 4/1 KD during chemo-radiation, followed by a modified Atkins diet during monthly chemotherapy. At the end of this period patients will follow a normal low carbohydrate diet similar to a Diabetic diet. The dietitian will follow the patient over the course of treatment. The patient will take and record ketone and glucose blood levels daily from start to end of treatment MRI scan, and meet with the dietitian weekly during radiation, at follow-up visits and on an as-needed basis.
Radiation: Radiation therapy — Patients receive standard dose (60Gy/30 fractions) external beam radiation
Drug: Temozolomide — patients receive standard dose (75 mg/kg/day) temozolomide by mouth daily with radiation for 6 weeks. patients will also have standard maintenance dose (150-200 mg/kg/day) for five days each month for 12 cycles following radiation course.
  Other Names: Temodar(R); chemotherapy

SUMMARY:
This study aims to see if reducing blood sugar and increasing ketones (a metabolic product that comes from using fats for energy) can increase survival and enhance the the effects of standard radiation and chemotherapy treatments used to treat glioblastoma multiforme (GBM). These changes occur from use of a ketogenic diet. This research has 2 goals:

1. Show that patients can tolerate the diet and maintain low blood glucose and high blood ketone levels.
2. Show if this diet enhances the effectiveness of standard treatment by prolonging survival of patients with a GBM.

DETAILED DESCRIPTION:
The investigators propose to offer this study to patients with newly diagnosed glioblastoma multiforme (GBM) that undergo gross total resection (GTR) or subtotal resection (STR) of their tumor. Post-operatively, these patients and their families will be instructed in the implementation of the Ketogenic Diet (KD) and it will be started as soon as possible following surgery to achieve ketosis and reduction of blood sugar. Patients will receive standard chemoradiotherapy with fractionated external beam radiation (60Gy) and concurrent oral temozolomide chemotherapy followed by 12 adjuvant cycles of temozolomide chemotherapy on a standard dose schedule. Outcome measures of the study group will be compared to historic controls in the treatment arm from the European Organization for Research and Treatment of Cancer (EORTC) temozolomide study published by Roger Stupp et al, New England Journal of Medicine, March 10, 2005.

Note: Gross Total Resection (GTR), Subtotal Resection (STR), temozolomide (Temodar), and radiation therapy are routine care for GBM and are not an investigational component of this study.

Study end-points:

Primary: Ketogenic diet (KD) tolerance and compliance in brain tumor patients. The diet will be considered tolerable if the patient chooses to remain compliant. Compliance is monitored by the dietician using self reporting of diet, blood glucose and blood ketone levels.

Secondary: Overall survival, time to recurrence, health and therapy-related quality of life. Overall survival and progression free survival will be measured and compared to the historic controls who received chemoradiotherapy in standard dose scheduling.

Laboratory correlate: Molecular/immunohistochemical analysis of tumors that do and do not respond to a KD.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, 18 - 80 years of age,
* a single enhancing lesion of the brain with MRI appearance consistent with GBM
* Pathologic confirmation of GBM
* Zubrod Performance Scale (ZPS) < 2
* Must be able to undergo MRI imaging with gadolinium
* Must have access to a computer and the internet (to use KetoCalculator© on-line Database)

Exclusion Criteria:

* unable to undergo MRI with gadolinium
* genetic disorders of fat metabolism
* patients receiving sodium valproate (may cause false ketone reading in urine)
* diabetes
* enrolled in another treatment trial for GBM

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-10 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 8 weeks
  Number of participants with adverse events from initiation of ketogenic diet through end of radiation (while on ketogenic diet)

SECONDARY OUTCOMES:
overall survival | 2 years
  overall survival
time to progression | 2 years
  time to progression
quality of life | 2 years
  patient reported outcome of their quality of life using FACT-BR (version 4) survey

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne C Scheck, PhD, Study Chair — Barrow Neurological Research
Locations (1):
- Barrow Neurological Institute at St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States

REFERENCES:
- [Background] Abdelwahab MG, Fenton KE, Preul MC, Rho JM, Lynch A, Stafford P, Scheck AC. The ketogenic diet is an effective adjuvant to radiation therapy for the treatment of malignant glioma. PLoS One. 2012;7(5):e36197. doi: 10.1371/journal.pone.0036197. Epub 2012 May 1. PMID 22563484
- [Background] Scheck AC, Abdelwahab MG, Fenton KE, Stafford P. The ketogenic diet for the treatment of glioma: insights from genetic profiling. Epilepsy Res. 2012 Jul;100(3):327-37. doi: 10.1016/j.eplepsyres.2011.09.022. Epub 2011 Oct 22. PMID 22019313
- [Background] Stafford P, Abdelwahab MG, Kim DY, Preul MC, Rho JM, Scheck AC. The ketogenic diet reverses gene expression patterns and reduces reactive oxygen species levels when used as an adjuvant therapy for glioma. Nutr Metab (Lond). 2010 Sep 10;7:74. doi: 10.1186/1743-7075-7-74. PMID 20831808